CLINICAL TRIAL: NCT00019357
Title: Cellular Immunotherapy With Autologous T Lymphocytes Stimulated With the Patient's Tumor-Specific Mutated Ras Peptides
Brief Title: Interleukin-2 Plus Activated White Blood Cells in Treating Patients With Cancer That Has Not Responded to Chemotherapy or Radiation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065811; NCI-97-C-0144; NCI-T97-0059; NCT00001583 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2004-04-22 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2001-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic autologous lymphocytes
Biological: therapeutic tumor infiltrating lymphocytes

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Combining white blood cells, which have been activated by a vaccine, with interleukin-2 may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-2 plus activated white blood cells in treating patients with cancer that has not responded to chemotherapy or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of expansion and the reinfusion of specific T-cell lines (peptide-specific activated lymphocytes), in combination with interleukin-2, in patients who were vaccinated with ras peptides. II. Assess immunologic status or antitumor response that may occur with this treatment in these patients.

OUTLINE: Autologous peptide-specific activated lymphocytes (PAL), previously harvested from the patient following vaccination on a different protocol, are expanded and reinfused intravenously; this is followed by a 4 hour observation period. Patients then receive interleukin-2 (IL-2) administered subcutaneously 5 days a week for 2 weeks; the first dose of IL-2 is administered at least 4 hours after PAL infusion. Patients are followed once a month for 2 months after treatment.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients must be enrolled to be treated with mutated ras peptides vaccine on another protocol Malignant disease for which no further chemotherapy or radiation options to increase survival are available No history of CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL SGOT or SGPT no greater than 4 times normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No active ischemic heart disease (i.e., NYHA class III or IV cardiac disease) No myocardial infarction within past 6 months No history of congestive heart failure No ventricular arrhythmias or other arrhythmias requiring therapy Other: HIV negative No hepatitis B or C infection No active infection requiring antibiotics No history of autoimmune disease (e.g., autoimmune neutropenia, thrombocytopenia, or hemolytic anemia; systemic lupus erythematosus, Sjogren syndrome, or scleroderma; myasthenia gravis; Goodpasture syndrome; Addison's disease, Hashimoto's thyroiditis, or active Graves' disease) No active second malignancy other than curatively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered Chemotherapy: At least 4 weeks since prior chemotherapy and recovered Endocrine therapy: At least 4 weeks since prior steroids and recovered No concurrent steroids Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Samir N. Khleif, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States